CLINICAL TRIAL: NCT05874258
Title: Improving Vision and Quality of Life in Patients With Glaucoma Using Non-invasive Brain Stimulation and Perceptual Learning: A Randomized Clinical Trial
Brief Title: Glaucoma Rehabilitation Using ElectricAI Transcranial Stimulation (GREAT) - Randomized Controlled Trial Using Combined Perceptual Learning and Transcranial Electrical Stimulation for Vision Enhancement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); University of Waterloo (Other); University of Magdeburg (Other)
Responsible Party: Principal Investigator, Allen MY Cheong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20190905001
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma
Keywords: glaucoma; transcranial direct current stimulation (tDCS); perceptual learning (PL)
MeSH Terms: conditions — Glaucoma | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: A prospective, double-masked, randomized, placebo-controlled training RCT design
Who Masked: Participant, Outcomes Assessor
Masking Description: Masked investigators responsible for all outcome measures and unmasked investigators responsible for group allocation and intervention. A set of random numbers will be generated by computer and the simple random sampling method (which matches according to age and gender) will be used to allocate the eligible participants into 3 groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real-PL + Real-tES (tDCS) (Experimental): Participant will receive 30 training sessions with real PL and real tES (tDCS): 3-4 sessions per week, about 1 hour per session
  Interventions: Other: Real-PL training + Real-tES(tDCS)
- Real-PL + Sham-tES (tDCS) (Experimental): Participant will receive 30 training sessions with real PL and sham tES (tDCS): 3-4 sessions per week, about 1 hour per session
  Interventions: Other: Real-PL training + Sham-tES (tDCS)
- Placebo-PL + Sham-tES (tDCS) (Placebo Comparator): Participant will receive 30 training sessions with placebo PL and sham tES (tDCS): 3-4 sessions per week , about 1 hour per session
  Interventions: Other: Placebo-PL training + Sham-tES (tDCS)

INTERVENTIONS:
Other: Real-PL training + Real-tES(tDCS) — PLtraining : around 40mins, tDCS: 20mins
  Arms: Real-PL + Real-tES (tDCS)
Other: Real-PL training + Sham-tES (tDCS) — PL training : around 40mins, tDCS: 20mins
  Arms: Real-PL + Sham-tES (tDCS)
Other: Placebo-PL training + Sham-tES (tDCS) — PL training : around 40mins, tDCS: 20mins
  Arms: Placebo-PL + Sham-tES (tDCS)

SUMMARY:
Glaucoma is a complex disease that can result in progressive vision loss. It is the second leading cause of blindness, accounting for 23% of permanent blindness in Hong Kong. There are no treatments that restore vision lost to glaucoma. However, recent studies have shown that vision can be improved by perceptual learning (PL) and transcranial electrical stimulation (tES). This study will examine the effect of perceptual learning and tES on improving quality of life, visual function and functional performance in patients with peripheral field loss due to glaucoma. It is phase 2 of Glaucoma Rehabilitation Using ElectricAI Transcranial Stimulation (GREAT) project.

DETAILED DESCRIPTION:
Study design:

This study uses a prospective, double-masked, randomized, placebo-controlled training RCT design.

The eligible participants will be randomly allocated into 3 groups:

(A) Placebo-Perceptual learning + Sham-tES; (B) Real-Perceptual learning + Sham-tES; (C) Real-Perceptual learning + Real-tES.

All participants will complete forty-three study visits:

Visit 1: Eligibility assessment (refer to the recruitment criteria); Visit 2-3: Outcome measures (Pre-intervention/ baseline); Visit 4-13: 10 sessions intervention (1st batch); Visit 14-15: Interim 1 Outcome measures; Visit 16-25: 10 sessions intervention (2nd batch); Visit 26-27: Interim 2 Outcome measures; Visit 28-37: 10 sessions intervention (3rd batch); Visit 38-39: Post-training 1 Outcome measures; Visit 40-41: Post-training 2 Outcome measures (to evaluate the retention effect after 1 month); Visit 42-43: Post-training 3 Outcome measures (to evaluate the retention effect after 2 months).

Six sessions of assessment will be conducted: (1) Baseline; (2) Interim-1 (after 10-sessions training); (3) Interim-2 (after 20-sessions training); (4) Post-1 (after 30-sessions training); (5) Post-2 (1-month post training); and (6) Post-3 (2-month post training).

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 80 years;
* Diagnosis of primary open angle or normal tension glaucoma with relative scotoma in both eyes;
* A relative scotoma defined as a Humphrey Field Analyser (HFA) threshold perimetry loss (mean deviation of -6dB) within the central 24 degree of the visual field for at least one eye;
* Best-corrected distance visual acuity of 6/12 or better (equivalent to 0.3 logMAR acuity or better to confirm that participant's central vision is preserved).
* Stable vision and visual field loss for at least 3 months;
* With a cognitive functional score of 22 or above in the Montreal Cognitive Assessment - Hong Kong version (HK-MoCA) (to confirm participant's intact cognitive function).

Exclusion Criteria:

* Ocular diseases other than glaucoma (e.g. age-related macular degeneration, diabetic retinopathy, moderate to severe cataract) or severe hearing impairment (to ensure that participant can hear the instructions clearly during assessments and training);
* Severe medical problems (e.g. stroke, Parkinson's disease) or self-reported neurological (e.g. brain surgery, brain tumor, peripheral neuropathy), or cognitive disorders (e.g. diagnosed dementia or cognitive impairment);
* Self-reported vestibular or cerebellar dysfunction, history of vertigo;
* Using any medications for any neurological conditions or psychiatric drugs (e.g. sedative, hypnotic) that might interfere motor control;
* Contraindications for non-invasive brain stimulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual field test | Change from baseline at 5weeks, change from baseline at 10weeks, change from baseline at 15weeks, change from baseline at 19weeks, changes from baseline at 23weeks
  Visual field test is measured monocularly using the 24-2 Swedish interactive threshold algorithm (SITA) standard tests by Humphrey Visual Field Analyzer (HFA, Carl Zeiss Meditec Inc., California). The mean deviation (MD), pattern standard deviation (PSD), and visual field index (VFI) are recorded and the MD of 24-2 visual field test is used as primary outcome of intervention effectiveness.

SECONDARY OUTCOMES:
High Resolution Perimetry (HRP) | Change from baseline at 5weeks, change from baseline at 10weeks, change from baseline at 15weeks, change from baseline at 19weeks, changes from baseline at 23weeks
  The current HRP is a valid and reliable computer-based visual field assessment based upon a previously well-established program. The revised HRP uses circular geometry instead of a rectangle to present stimuli, while maintaining its high-resolution advantage. During the HRP test, suprathreshold stimuli are presented in a radial pattern within 20 degrees, with a step size of 3 degrees. These stimuli are presented monocularly at a total of 98 positions, with the order of presentation randomized. To ensure a stable result and accurate assessment of participants' responses, the HRP test is repeated five times. Throughout the HRP test, fixation is monitored by an infrared eye tracker (SR Research, Eyelink Portable Duo).
Electroencephalography (EEG) | Change from baseline at 15weeks, change from baseline at 19weeks, changes from baseline at 23weeks
  64-channel electroencephalography(EEG) recordings from Neuroscan will be used to understand the electrophysiological changes in the intervention. A standard visual evoked potential task (VEP) and a specific designed SSVEP task will be used to assess the functional integrity of central vision and peripheral function. Besides, resting-state EEG will be recorded to measure the functional connectivity at different timepoints. ERP components (such as P100, N1 and N2) in VEP, tagging frequency response in SSVEP, and the power correlation in resting state will be analyzed as physiological indicators.
Gait Test | Change from baseline at 15weeks, change from baseline at 19weeks, changes from baseline at 23weeks
  All participants will be asked to walk along a 7-m walkway at their normal pace. Two disturbing factors will be introduced while walking: visual searching task and obstacle crossing. For trials with visual search, visual stimuli will be presented on the monitor (located at the end of the walkway) when the participant crosses the obstacle. For trials with obstacle crossing, an obstacle with two different colors (grey for low contrast and yellow for high contrast obstacle) of two different heights (2.5x60x5 cm or 2.5x60x15 cm) are positioned at the middle of the walkway. Participants' gait parameters including hip flexion/extension (degree), knee Min/Max (degree), ankle flexion/extension (degree), head flexion/extension (degree), walking speed (mm/s), step width (mm), and toe clearance(mm) will be measured and analyzed for each condition.
Balance function | Change from baseline at 5weeks, change from baseline at 10weeks, change from baseline at 15weeks, change from baseline at 19weeks, changes from baseline at 23weeks
  Balance function will be evaluated for the following two conditions:
  1. Static Balance: Participants will be asked to stand on a force place with a foam while performing visual searching. Parameters including maximum antero-posterior amplitude (mm), maximum medio-lateral amplitude (mm), total sway path (mm), and root mean square sway (mm/s) will be analyzed.
  2. Perturbed Balance: Participants will be asked to stand on a force place which will translate forward or backward while performing visual searching. Parameters including latency (ms) reacting to the perturbation, maximum antero-posterior amplitude (mm), maximum medio-lateral amplitude (mm), total sway path (mm), and root mean square sway (mm/s) will be analyzed.
Questionnaires for QoL | Change from baseline at 15weeks, change from baseline at 19weeks, changes from baseline at 23weeks
  National Eye Institute Visual Function Questionnaire 25 (NEI-VFQ 25) and Low Vision Quality of Life (LVQoL) will be used to evaluate the patient-perceived outcome of the intervention on daily living. In NEI-VFQ 25, more positive person measures indicates greater visual ability, and more negative person measures have less visual ability. In the LVQoL, the completion results in a summed score between 0 (a low quality of life) and 125 (a high quality of life).

OTHER OUTCOMES:
Magnetic resonance spectroscopy (Optional) | Change from baseline at 15 weeks
  Magnetic resonance spectroscopy (MRS) is a non-invasive imaging technique that can be used to study the chemical composition of tissues, including the brain. Changes in GABAergic and Glutamatergic concentrations within the MRS voxels will be used to evaluate the mechanistic changes in the brain. To study the mechanism of glaucoma, we plan to use MEGA-PRESS in primary visual cortex(V1) of the brain to understand the neural and metabolic mechanisms.
BDNF concentration in serum and tears (Optional) | Change from baseline at 15 weeks
  Serum BDNF concentration will be measured using an enzyme-linked immunoassay (ELISA) kit and liquid chromatography-mass spectrometry(LCMS). DNA will be extracted from the leucocytes for the determination of BDNF Val66Met polymorphism (rs6265G>A) using a method based on polymerase chain reaction (PCR).
  Collection of tear sample by capillary tube (10 ul) or Schirmer Strip in labelled eppendorf tube and keep them frozen immediately. Tear BDNF concentration will be measured using an enzyme-linked immunoassay (ELISA) kit and liquid chromatography-mass spectrometry.
Cortisol concentration in serum and tears (Optional) | Change from baseline at 15 weeks
  Cortisol concentration will be measured using an enzyme-linked immunoassay (ELISA) kit and liquid chromatography-mass spectrometry(LCMS).
  Collection of tear sample by capillary tube (10 ul) or Schirmer Strip in labelled eppendorf tube and keep them frozen immediately. Tear Cortisol concentration will be measured using an enzyme-linked immunoassay (ELISA) kit and liquid chromatography-mass spectrometry.
Questionnaire of psychological state | Change from baseline at 15weeks, change from baseline at 19weeks, change from baseline at 23weeks.
  Perceived Stress Scale (PSS-10) and Patient Health Questionnaire - 9 (PHQ9) will be used to evaluated the stress and depression severity of the outcome of the intervention of participant. Individual scores on the PSS-10 can range from 0 to 40 with higher scores indicating higher perceived stress. In PHQ9, the completion results in a summed score between 0 (none minimal) to 27 (severe).
Questionnaire of fear of falling | Change from baseline at 15weeks, change from baseline at 19weeks, change from baseline at 23weeks.
  Falling is a significant concern for glaucoma patients, with the fear of falling being a major contributing factor to the incidence of falls. Moreover, fear of falling is associated with a decreased physical and social activity. The Chinese version of the Falls Efficacy Scale- International (FES-I) is a validated and reliable questionnaire used to assess fear of falling in everyday life. This questionnaire includes sixteen items that are related to common daily activities, each graded on a scale of from 1 (not at all concerned) to 4 (very concerned). Higher scores indicate a greater concern about falling, which may indicate a poorer balance ability.
Kinetic visual field | Change from baseline at 15weeks, change from baseline at 19weeks, change from baseline at 23weeks.
  The kinetic test is highly sensitive in detecting changes in the far peripheral visual field, which significantly correlates with balance function and gait performance. The binocular kinetic visual field is measured using Octopus 900 perimetry (Haag-Streit AG, Switzerland). Tests are done in the kinetic mode using the standard protocol (sixteen vectors), with a stimulus size of III4e moving at a speed of 5 degrees/sec to map the hill of vision. Any changes in the area of the isopter over time would indicate the effect of training on the kinetic visual field.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: available: 3mths after data complication
Access Criteria: The requestor's affiliation and purpose are required to get the access.

REFERENCES:
- [Derived] Jia S, Mei X, Chen L, Chan LH, Tsang C, Suen V, Li T, Zaw MW, Liu A, Thompson B, Sabel B, Woo G, Leung CKS, Yip SP, Chang DHF, Cheong AMY. Glaucoma Rehabilitation using ElectricAI Transcranial Stimulation (GREAT)-study protocol for randomized controlled trial using combined perceptual learning and transcranial electrical stimulation for vision enhancement. Trials. 2024 Jul 22;25(1):501. doi: 10.1186/s13063-024-08314-3. PMID 39039582